CLINICAL TRIAL: NCT05349682
Title: Transcatheter Geniculate Arterial Embolization: Treatment and Monitoring of Response
Brief Title: Bayer OA Knee Pain Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00113621
Record Dates: First submitted 2022-03-28; First posted 2022-04-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GAE and MRI treatment arm (Experimental): GAE is geniculate artery embolization.
  Interventions: Diagnostic Test: dynamic contrast enhanced MRI; Procedure: geniculate artery embolization

INTERVENTIONS:
Diagnostic Test: dynamic contrast enhanced MRI — An MRI study of the knee will be done to check the degree of osteoarthritis and blood flow to the affected knee. This scan will take about 1-2 hour(s).
Procedure: geniculate artery embolization — The physician will perform a diagnostic angiography, where they will take pictures of vessels near the knee that will be treated. Once the artery to be treated is identified, the doctor will guide a thin wire called a microwire, and a plastic tube called a microcatheter to the targeted artery, and more pictures of vessels at the knee will be taken. This picture will be used to see if there are any abnormal vessels at the knee, such as abnormal blood flow, abnormal vessel connections (between the veins and arteries), or new blood vessel growth. Once the targeted artery at the knee is confirmed, the doctor will inject enough particle embolic (Embozene) to slow or stop the blood flow in the geniculate artery. Once all vessels are treated, a final angiogram (pictures of blood vessels) will be performed to ensure that the blood flow has slowed.

SUMMARY:
The objective of this study is to investigate if MRI can be used to evaluated effect of knee artery embolization for knee osteoarthritis. Participants be evaluated in clinic, obtain a knee MRI, undergo embolization of the symptomatic knee, and follow up in clinic at 1, 6, and 12 months after embolization. A second MRI is obtained 6 months after embolization. Participants will keep a record of their pain level and treatment and answer questionnaires at each visit.

In addition, this study aims to determine the effects of knee artery embolization on the amount of opioid (pain reliever drugs) needed to manage osteoarthritis-associated pain and change in quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 to 90
2. Symptomatic osteoarthritis of one or both knees, with Kellgren-Lawrence grade 1-3 assessed by weight-bearing knee radiography, including post-traumatic osteoarthritis
3. One or more months of non-surgical therapy for knee pain such as joint injections, oral NSAIDs, or opioid analgesia
4. Subjects able to provide informed consent. As this is a study of pain, patients must be able to consent for themselves.
5. Patients without contraindication to MRI imaging with gadolinium-based contrast.

Exclusion Criteria:

1. Anaphylaxis to gadolinium or iodinated contrast media
2. Impaired renal function with GFR <30ml/min
3. Severe atherosclerotic disease of the lower extremity precluding percutaneous angiographic access to the involved geniculate artery(ies)
4. Active septic arthritis of the symptomatic knee within 2 months of screening
5. Malignancy of the involved knee
6. Rheumatoid Arthritis or Gout
7. Prior knee surgery
8. Hemarthrosis
9. Females who are pregnant or plan to become pregnant during the study. All participants able to become pregnant will be administered a urine pregnancy test.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in enhancement time intensity curves obtained from CE-MRI | change from baseline at 6 month post procedure
  To evaluate the effects of particle embolization on knee osteoarthritis progression using enhancement time intensity curves obtained from CE-MRI (Contrast Enhanced Magnetic Resonance Imaging)
Change in Whole-Organ Magnetic Resonance Scoring (WORMS) | change from baseline at 6 month post procedure
  To evaluate the effects of particle embolization on knee osteoarthritis progression using the WORMS scoring system. The higher the score, the worse the OA is. The scoring ranges from 0-332.
Change in Multicenter Osteoarthritis Study (MOST) grading system for synovitis | change from baseline at 6 month post procedure
  To evaluate the effects of particle embolization on knee osteoarthritis progression using the MOST grading system for synovitis. The higher the score, the worse the synovial inflammation is. The scoring ranges from 0-13. 0-4 normal or equivocal synovitis, 5-8 mild synovitis, 9-12 moderate synovitis, and 13 or greater is severe synovitis.
Number of participants with 50% reduction in pain scores | change from baseline at 1 month post procedure
  To determine the effects of geniculate artery embolization (GAE) on opioid requirements for managing OA associated pain. Assess pain using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Knee Injury and Osteoarthritis Outcome Score (KOOS). WOMAC is scored from 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. Higher scores indicate worse pain, stiffness, and function limitation. KOOS score is from 0-100, 0 being extreme problems and 100 being no problems.
Number of participants with 50% reduction in pain scores | change from baseline at 6 month post procedure
  To determine the effects of geniculate artery embolization (GAE) on opioid requirements for managing OA associated pain. Assess pain using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Knee Injury and Osteoarthritis Outcome Score (KOOS). WOMAC is scored from 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. Higher scores indicate worse pain, stiffness, and function limitation. KOOS score is from 0-100, 0 being extreme problems and 100 being no problems.
Number of participants with 50% reduction in pain scores | change from baseline at 12 month post procedure
  To determine the effects of geniculate artery embolization (GAE) on opioid requirements for managing OA associated pain. Assess pain using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Knee Injury and Osteoarthritis Outcome Score (KOOS). WOMAC is scored from 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. Higher scores indicate worse pain, stiffness, and function limitation. KOOS score is from 0-100, 0 being extreme problems and 100 being no problems.
Incidence of adverse events associated with GAE | 1 month post procedure
  The number of adverse events per participant
Incidence of adverse events associated with GAE | 6 month post procedure
  The number of adverse events per participant
Incidence of adverse events associated with GAE | 12 month post procedure
  The number of adverse events per participant

CONTACTS AND LOCATIONS:
Overall Officials: Andre Uflacker, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share anonymized DCE-MRI data with consulting radiologists.
Time Frame: duration of the study
Access Criteria: The data will only be shared via encrypted email or encrypted cloud repository.